CLINICAL TRIAL: NCT01733706
Title: Evaluation of Early Smoking Reduction or Cessation by Means of no Nicotine Electronic Cigarette Added to Standard Counselling.
Brief Title: Early Smoking Reduction or Cessation by Means of no Nicotine Electronic Cigarette Added to Standard Counselling.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO S617/211
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2015-12

CONDITIONS: Cancer; Myocardial Infarction
Keywords: No Nicotine Electronic Cigarette; Antismoke intervention
MeSH Terms: conditions — Neoplasms; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard counseling (Active Comparator): a psychologist will provide standard counseling
  Interventions: Other: Standard counseling
- No nicotine electronic cigarette (Experimental): patients will receive standard counseling as well as an electronic cigarette
  Interventions: Device: No nicotine electronic cigarette; Other: Standard counseling

INTERVENTIONS:
Device: No nicotine electronic cigarette — The e-cigarette "T-FUMOTM" is a no nicotine electronic cigarette specifically designed to inactivate the early effects of the cessation of cigarette smoking, such as the craving caused by psychological reasons. It's formed by a filter which contains distilled water and food flavorings, an atomizer and a battery. On the opposite end to the filter there is a diode that lights up during aspiration. During the suction is generated hot air which, in contact with the liquid of the filter, generates steam which simulates the smoke of a traditional cigarette. The smoker has the sensation of smoking, but he does not suck the carcinogenic substances in traditional cigarettes and he does not assimilate nicotine.
  Other Names: e-cigarette "T-FUMOTM"
  Arms: No nicotine electronic cigarette
Other: Standard counseling — standard counseling

SUMMARY:
The aim of this study is the evaluation of early smoking reduction or cessation by means of no nicotine electronic cigarette added to standard counselling.

DETAILED DESCRIPTION:
Cigarette smoking is one of the major health problems in the modern world for the impact on morbidity and mortality with devastating effects on cardio-cerebrovascular system and on tumor onset. After years of scientific doubts, today the scientific world agrees to define cigarette smoking not a "vice" but a disease.

The aim is to evaluate the effect of no nicotine electronic cigarette use in patients with cancer or myocardial infarction, smoking at least 10 cigarettes per day for at least 10 years, in addition to counselling activity performed by specialised dedicated medical doctors.

If patient is eligible for this trial, he will be enrolled in this trial and randomized. Randomization will be performed using a web-based procedure. Study participants will be randomized to electronic cigarette added to standard counselling or only standard counselling. A calendar will be given to the patient to remember the dates of visits or telephone counselling. After the first visit patient will be followed every ten days for the first two month through outpatient clinic visits and telephone counselling. After the first two months patient will return at institute for a last outpatient clinic visit at sixth month.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of cancer and recently operated at European Institute of Oncology at Milan (Italy);
* patients with a diagnosis of hematology cancer treated at Foundation "San Raffaele del Monte Tabor" at Milan;
* patient with a recent occurrence of acute myocardial infarction from Monzino Cardiology Centre at Milan;
* age greater than 18 years;
* smokers stable for at least 10 cigarettes per day for at least 10 years.

Exclusion Criteria:

* patients with life expectancy less than 6 months;
* patients who have undertaken structured attempts to stop smoking over the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked | two months after event (cancer or myocardial infarction)
psychological conditions | two months after event (cancer or myocardial infarction)
  psychological conditions will be assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cipolla, MD, Study Chair — European Institute of Oncology
Locations (2):
- Italy (2):
  - European Institute of Oncology, Milan
  - Istituto Scientifico San Raffaele del Monte Tabor IRCCS, Milan